CLINICAL TRIAL: NCT04647643
Title: Real-World Safety Analysis of Paclitaxel Devices Used for the Treatment of Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: Lahey Clinic (Other)
Collaborators: National Evaluation System for health Technology Coordinating Center (Other); Society for Vascular Surgery Patient Safety Organization (Other)
Responsible Party: Principal Investigator, Sourbha Dani, Staff Cardiologist, Lahey Clinic
Other Study IDs: 20203069FH; 6292-2020-2AS-1001-Phase1 (Other Grant/Funding Number: NESTcc)
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paclitaxel Drug Coated Balloon: Patients treated with paclitaxel drug-coated balloon
  Interventions: Drug: Paclitaxel
- Paclitaxel Drug Coated Stent: Patients treated with paclitaxel drug-coated stent
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel to treat peripheral arterial disease
  Other Names: Taxol

SUMMARY:
Treatment with paclitaxel-based endovascular devices (PED) has become a common treatment option for patients with peripheral artery disease (PAD) involving the femoral-popliteal artery. However, an aggregate level meta-analysis identified an association between the use of PED and increased all-cause mortality at both two and five-year follow-up intervals, though there are significant limitations of these analyses. Exploration of real-world data has been suggested as a means to further investigate the safety of PED. The current study explores the association of PED and mortality in real-world data using U.S. commercial claims from the FAIR Health data warehouse.

DETAILED DESCRIPTION:
Treatment with paclitaxel-based endovascular devices (PED) has become a common treatment option for patients with peripheral artery disease (PAD) involving the femoral-popliteal artery. However, an aggregate level meta-analysis identified an association between the use of PED and increased all-cause mortality at both two and five-year follow-up intervals, though there are significant limitations of these analyses. Exploration of real-world data has been suggested as a means to further investigate the safety of PED. The current study explores the association of PED and mortality in real-world data using U.S. commercial claims from the FAIR Health data warehouse.

This study aims to evaluate the relative safety of paclitaxel used as an antiproliferative agent in the treatment of symptomatic PAD in a real-world scenario. We will analyze Paclitaxel Drug-Coated Balloons (DCB) and Paclitaxel Drug-Eluting Stents (DES), in aggregate and as unique exposures using propensity score-matched survival analysis. (Inverse probability of Treatment Weighting).

Commercial claims of patients who underwent endovascular interventional treatment of the femoral or popliteal arteries for symptomatic PAD between 1/1/15 and 12/31/2019 will form the study population. Three separate safety analyses will be performed. 1. Paclitaxel Drug coated balloons (DCB) as compared with propensity-matched patients treated with plain transluminal balloon angioplasty (PTA). 2. Paclitaxel delivering Drug-Eluting Stents (DES) as compared with propensity-matched cases using bare-metal stents (BMS). 3. Patients treated with either paclitaxel DCB or paclitaxel DES (any PTX) compared with propensity-matched controls (non-PTX,with DCB patients, matched to patients treated with PTA, and DES patients matched to patients treated with BMS).

All proposed analyses will be performed using R 4.01 implemented within the DELTA analytic engine. DELTA is an active surveillance safety system that can monitor clinical data repositories for safety signals and has been validated to support risk-adjusted prospective safety surveillance analyses of complex clinical datasets.

ELIGIBILITY:
Inclusion Criteria:

* All patients, age 18 or older, who had a health insurance claim for outpatient endovascular treatment of the femoral or popliteal arteries for symptomatic PAD will be included. The diagnosis and treatment of PAD in the femoral and popliteal arteries will be identified by CPT/HCPCS and ICD-9 and ICD-10 PCS codes.
* Presence of at least one additional outpatient or inpatient claims, at least 12 months following the index procedure, in order to demonstrate continued enrollment in health insurance coverage.

Exclusion Criteria:

* Age <18 years
* No qualifying peripheral arterial endovascular procedure
* Inpatient procedure
* Patients without any linked claim record more than 12 months after the index procedure, not known to have died or entered hospice care within the first 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial claims of patients who underwent endovascular interventional treatment of the femoral or popliteal arteries for symptomatic PAD between 1/1/15 and 12/31/2019 will form the study population. Three separate safety analyses will be performed. 1. Paclitaxel Drug coated balloons (DCB) as compared with propensity-matched patients treated with plain transluminal balloon angioplasty (PTA). 2. Paclitaxel delivering Drug-Eluting Stents (DES) as compared with propensity-matched cases using bare-metal stents (BMS). 3. Patients treated with either paclitaxel DCB or paclitaxel DES (any PTX) compared with propensity-matched controls (non-PTX,with DCB patients, matched to patients treated with PTA, and DES patients matched to patients treated with BMS).
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Survival | 4 years post intervention
  Freedom from death of any cause

SECONDARY OUTCOMES:
Survival | 2 years post intervention
  Freedom from death of any cause
Retreatment | 2 years post intervention
  Retreatment with repeat revascularization (open or endovascular)
Amputation | 2 years post intervention
  Freedom from amputation

OTHER OUTCOMES:
Survival for age groups | 4 years and 2 years post intervention
  Freedom from death in the age groups 18-34, 35-44, 45-54, 55-64, 65-74, 75 and above
Survival for demographics and special baseline variables | 4 years and 2 years post intervention
  Freedom from death in females, patients with claudication, CKD and dialysis, history of CAD, history of cancer
Survival for special treatment category | 4 years and 2 years post intervention
  Freedom from death in patients with patients receiving paclitaxel-coated device as a second procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sourbha S Dani, MD, MSc, Principal Investigator — Lahey Hospital & Medical Center; Frederic S Resnic, MD, MSc, Study Director — Lahey Hospital & Medical Center; Robbert Zusterzeel, MD, MPH, PhD, Study Chair — NESTcc
Locations (1):
- Lahey Clinic, Inc, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Zeller T, Roubin GS, Burket MW, Khatib Y, Snyder SA, Ragheb AO, White JK, Machan LS; Zilver PTX Investigators. Paclitaxel-eluting stents show superiority to balloon angioplasty and bare metal stents in femoropopliteal disease: twelve-month Zilver PTX randomized study results. Circ Cardiovasc Interv. 2011 Oct 1;4(5):495-504. doi: 10.1161/CIRCINTERVENTIONS.111.962324. Epub 2011 Sep 27. PMID 21953370
- [Result] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Snyder SA, O'Leary EE, Tepe G, Scheinert D, Zeller T; Zilver PTX Investigators. Sustained safety and effectiveness of paclitaxel-eluting stents for femoropopliteal lesions: 2-year follow-up from the Zilver PTX randomized and single-arm clinical studies. J Am Coll Cardiol. 2013 Jun 18;61(24):2417-2427. doi: 10.1016/j.jacc.2013.03.034. Epub 2013 Apr 10. PMID 23583245
- [Result] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254
- [Result] Rocha-Singh KJ, Duval S, Jaff MR, Schneider PA, Ansel GM, Lyden SP, Mullin CM, Ioannidis JPA, Misra S, Tzafriri AR, Edelman ER, Granada JF, White CJ, Beckman JA; VIVA Physicians, Inc. Mortality and Paclitaxel-Coated Devices: An Individual Patient Data Meta-Analysis. Circulation. 2020 Jun 9;141(23):1859-1869. doi: 10.1161/CIRCULATIONAHA.119.044697. Epub 2020 May 6. PMID 32370548
- [Result] Secemsky EA, Kundi H, Weinberg I, Jaff MR, Krawisz A, Parikh SA, Beckman JA, Mustapha J, Rosenfield K, Yeh RW. Association of Survival With Femoropopliteal Artery Revascularization With Drug-Coated Devices. JAMA Cardiol. 2019 Apr 1;4(4):332-340. doi: 10.1001/jamacardio.2019.0325. PMID 30747949
- [Result] Secemsky EA, Kundi H, Weinberg I, Schermerhorn M, Beckman JA, Parikh SA, Jaff MR, Mustapha J, Rosenfield K, Yeh RW. Drug-Eluting Stent Implantation and Long-Term Survival Following Peripheral Artery Revascularization. J Am Coll Cardiol. 2019 May 28;73(20):2636-2638. doi: 10.1016/j.jacc.2019.02.020. Epub 2019 Mar 1. No abstract available. PMID 30831175
- [Result] Behrendt CA, Sedrakyan A, Peters F, Kreutzburg T, Schermerhorn M, Bertges DJ, Larena-Avellaneda A, L'Hoest H, Kolbel T, Debus ES. Editor's Choice - Long Term Survival after Femoropopliteal Artery Revascularisation with Paclitaxel Coated Devices: A Propensity Score Matched Cohort Analysis. Eur J Vasc Endovasc Surg. 2020 Apr;59(4):587-596. doi: 10.1016/j.ejvs.2019.12.034. Epub 2020 Jan 8. PMID 31926836
- [Result] Resnic FS, Gross TP, Marinac-Dabic D, Loyo-Berrios N, Donnelly S, Normand SL, Matheny ME. Automated surveillance to detect postprocedure safety signals of approved cardiovascular devices. JAMA. 2010 Nov 10;304(18):2019-27. doi: 10.1001/jama.2010.1633. PMID 21063011
- [Result] Kumar A, Matheny ME, Ho KK, Yeh RW, Piemonte TC, Waldman H, Shah PB, Cope R, Normand SL, Donnelly S, Robbins S, Resnic FS. The data extraction and longitudinal trend analysis network study of distributed automated postmarket cardiovascular device safety surveillance. Circ Cardiovasc Qual Outcomes. 2015 Jan;8(1):38-46. doi: 10.1161/CIRCOUTCOMES.114.001123. Epub 2014 Dec 9. PMID 25491915
- [Result] Resnic FS, Majithia A. Registry-Based Surveillance of Medical-Device Safety. N Engl J Med. 2017 May 18;376(20):1995. doi: 10.1056/NEJMc1704006. No abstract available. PMID 28514621
- [Result] Hsieh FY, Lavori PW, Cohen HJ, Feussner JR. An overview of variance inflation factors for sample-size calculation. Eval Health Prof. 2003 Sep;26(3):239-57. doi: 10.1177/0163278703255230. PMID 12971199
- [Result] Vidi VD, Matheny ME, Resnic FS. Post-marketing device safety surveillance. Contemp Clin Trials. 2011 May;32(3):307-8. doi: 10.1016/j.cct.2011.02.002. Epub 2011 Feb 28. No abstract available. PMID 21371573
- [Result] Austin PC. Optimal caliper widths for propensity-score matching when estimating differences in means and differences in proportions in observational studies. Pharm Stat. 2011 Mar-Apr;10(2):150-61. doi: 10.1002/pst.433. PMID 20925139
- See also: McKeown L. Two trials halted in wake of study linking paclitaxel-coated devices to deaths in PAD — https://www.tctmd.com/news/two-trials-halted-wake-study-linking-paclitaxel-coated-devices-deaths-pad